CLINICAL TRIAL: NCT06239077
Title: Identifai Genetics Analytical Validation Study
Brief Title: Identifai Genetics Analytic Validity Study - Compound Heterozygosity and Samples Collection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Identifai Genetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL001
Record Dates: First submitted 2023-12-20; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-12

CONDITIONS: Prenatal Diagnosis; Genetics
Keywords: NIPS; NIPT

STUDY DESIGN:
Masking Description: Patient information is confidential and shared exclusively with the treating physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Identifai Genetics Analytic Validity - Compound Heterozygosity and Samples Collection (Experimental)
  Interventions: Other: Non Invasive Prenatal Test via blood sample

INTERVENTIONS:
Other: Non Invasive Prenatal Test via blood sample — Maternal - blood draw, Paternal - blood draw/Saliva sample

SUMMARY:
The purpose of this study is to validate a noninvasive prenatal diagnosis procedure for genetic conditions in the developing fetus by analyzing fetal genetic material present in the pregnant mother's blood.

DETAILED DESCRIPTION:
Amniocentesis (drawing fluid from inside the womb) and chorionic villus sampling (removing a very small amount of the developing placenta) are the current "gold standard" for diagnosis of genetic abnormalities in the developing fetus (unborn child) during the pregnancy. However, these procedures have small risks of miscarriage and are normally used for women with known risk factors for a genetic condition in the fetus. Finding a method to detect genetic changes in a fetus without performing a procedure associated with a risk for miscarriage may be helpful for the clinical care of pregnant patients in collaboration with their providers in the future.

It has been demonstrated that cell-free fetal (cff) DNA is present in the mother's bloodstream. This is already used to detect common conditions like Down Syndrome, a condition that all pregnancies are at risk for. The existing cffDNA tests are not currently able to detect if a fetus is a carrier or affected with the conditions parents are commonly screened for using carrier screening and other genomic tests. The study aim to test the use of new genetic techniques on cffDNA that can find if a fetus is affected with condition that one or both parents are carriers for. The study also aim to investigate if these new tools can detect other spontaneous and inherited genetic changes. This will make prenatal detection possible of many more genetic disorders than can currently be done by drawing blood from the mother. The Maternal and Paternal blood samples will be also used for the development of new methods to detect genetic abnormalities in the developing fetus.

ELIGIBILITY:
Inclusion Criteria:

General:

* Parental age≥18
* Singleton pregnancy
* Willingness and ability to provide informed consent to participate in study
* Patient having a diagnostic procedure (CVS, amniocentesis, cordocentesis) or delivering on site (obtain cord blood/cord segment)

Main Study:

* Gestational age: 10-23 weeks
* Parents are both carriers of different known pathogenic SNVs or short indels (<=5bp) in the same gene (compound heterozygosity).

Substudy:

* Gestational age ≥10 weeks
* Either parent or both carry a known structural variant and/or other chromosomal anomalies AND/OR Ultrasound highly suggestive of an underlying genetic aberration (e.g., cardiac outlet and 22q)

Exclusion Criteria:

* Any Multiple gestation is excluded (MCDA, DCDA, triplets, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women and father are recruited
Enrollment: 100 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analytic Validity - Sensitivity | 10 weeks
  The ability to correctly detect pregnancies that are positive for the suspected genetic condition arising from a compound heterozygosity scenario. It is calculated by assessing the proportion of true positive results among all pregnancies that actually have the condition. This calculation involves dividing the number of true positive cases by the total number of cases that truly have the condition (sum of true positive and false negative cases), thus providing a measure of the test's accuracy in correctly identifying the condition when it is actually present.
Analytic Validity - Specificity | 10 weeks
  The ability to accurately identify pregnancies that do not have the suspected genetic aberration arising from a compound heterozygosity scenario. It is calculated by determining the proportion of true negative results among all cases that are actually free from the condition. This involves dividing the number of true negative cases by the sum of true negative and false positive cases, providing a measure of the test's accuracy in correctly ruling out the condition in unaffected pregnancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No